CLINICAL TRIAL: NCT01652001
Title: Effectiveness of Malic Acid 1% in Patients With Xerostomia Induced by Drugs. Determination of Salivary Mucins and Buffering Capacity
Brief Title: Drug-induced Xerostomia. Evaluation of Malic Acid 1%, Salivary Mucins and Buffering Capacity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Gerardo Gomez Moreno, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Xerostomia-2012; PI10/00932 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2012-07-20; First posted 2012-07-27 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Xerostomia; Depression; Hypertension
Keywords: Xerostomia; Antidepressant agents; Antihypertensive agents
MeSH Terms: conditions — Xerostomia; Depression; Hypertension | interventions — malic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Malic Acid 1% (Experimental): Intervention group subjects was the delivery to the patients of a topical sialogogue, containing 1% malic acid, xylitol 10% and fluoride 0.05%(Xeros Dentaid Spray©, Dentaid, Barcelona, Spain).
  Spray was transferred by foreign personnel into identical opaque flasks(without any brand name)labeled A.
  Interventions: Drug: Malic Acid
- Control (Placebo Comparator): Control group was given a placebo with opaque flask(without any brand name)labeled B and with the same presentation and composition than Experimental group (excepting 1% malic acid).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Malic Acid — Oral spray for application into the oral cavity
  Other Names: XerosDentaid Spray; Flask labeled A
  Arms: Malic Acid 1%
Other: Placebo — Oral spray for application into the oral cavity
  Other Names: Flask labeled B
  Arms: Control

SUMMARY:
The aim of our study was to evaluate the clinical efficacy of a topical sialogogue spray containing 1% malic acid on patients affected by xerostomia caused by drugs.

This research took the form of a double-blind, randomized clinical trial at Faculty of Dentistry of University of Granada (Spain). Participants with antidepressant-induced and antihypertensive-induce xerostomia were divided into two groups: for the first 'intervention group' a topical sialogogue spray (1% malic acid) was applied, while for the second 'control group', a placebo spray was applied; for both groups the sprays were applied on demand during two weeks. The Dry Mouth Questionnaire (DMQ) was used to evaluate xerostomia levels before and after product/placebo application. Unstimulated and stimulated salivary flows rates, before and after application, were measured.

DETAILED DESCRIPTION:
- Patients and study Design The study was approved by the University of Granada Research Ethics Committee (Spain). All measurements and interventions were undertaken with the understanding and written consent of each participant according to Helsinki II Agreement.The study was designed as a double-blind randomized clinical trial following guidelines established by The Consort Statement (http://www.consort-statement.org/consort-statement/). All study participants were recruited from the Faculty of Dentistry of the University of Granada (Spain)at Drug Interactions in Dentistry clinical practice, between September and December 2011. Recruitment was supervised by research assistants.

All participants had a full medical history and saliva samples were collected at the Faculty of Dentistry of University of Granada (Spain) at the Pharmacological Investigation in Dentistry Research Group laboratory (CTS-654).

Sample size determination was based on the standard deviation of the main variable: the Dry Mouth Questionnaire (DMQ)was tested to determine the minimum sample size necessary to reliably confirm the hypothesis that a topical 1% malic acid sialogogue spray, combined with xylitol and fluoride, is effective for the treatment of xerostomia induced by antidepressant drugs over a two-week period. DMQ and saliva collection were measured the same day and by the same investigator.

* Clinical Intervention Once the participants had signed the informed consent form and anamnesis had been carried out, the following question was asked to every patient: "How often do you feel dry mouth?" Available answers were: "never", "sometimes", "usually" or "always." Those who answered "usually" or "always" were considered as suffering from xerostomia. Our clinical intervention among the intervention group subjects was the delivery to the patients of a topical sialogogue, containing 1% malic acid, xylitol 10% and fluoride0.05%(Xeros Dentaid Spray©, Dentaid, Barcelona, Spain) for two weeks, whereas a control group was given a placebo with the same presentation and composition (excepting 1% malic acid). Randomization was performed using the website http://www.randomization.com, obtaining a randomization plan, which assigned participants to either the intervention group or the control group. This randomization plan was delivered to a person unrelated to the study in order to prevent both participants and researchers from identifying the product.Both sprays were transferred by foreign personnel into two identical opaque flasks(without any brand name)labeled A and B containing respectively, either 1% malic acid or placebo.A code for randomization was kept in an opaque envelope in a safe environment and opened only at the end of the study. Data were analyzed by a third party blinded to the allocation results. 1% malic acid/placebo sprays were applied on demand, with a maximum of eight doses per day. No participants left the trial.
* Dry Mouth Questionnaire (DMQ) The DMQ, developed by Vissink et al., Gravenmade et al., van der Reijden et al. and Regelink et al. was used in order to obtain subjective information about the severity of xerostomia before and after treatment with malic acid/placebo. Every participant answered an initial questionnaire (DMQ 1) about the symptoms related to oral dryness, before receiving a spray (1% malic acid or placebo). After two weeks of applications, patients had to answer DMQ 1 again as well as an additional questionnaire (DMQ 2) about the efficacy of the sprays. Increased DMQ scores indicate improvement of xerostomia. DMQ 1 was used to assess the initial severity of oral dryness and in particular its impact on oral function: problems when chewing, swallowing, speaking and general impact on daily life.

DMQ 1 used a 0-to-4 rating scale where 0 = "very dry" and 4 = "not dry at all." After two weeks of treatment, DMQ 1 was repeated. DMQ 2 was designed to assess the impact of the spray on the symptoms of xerostomia, and was also based on a 0-to-4 rating scale where 0 = frequent restriction of oral function and 4= no restriction of oral function/no feeling of oral dryness. The effect of the frequency and duration of spray applications in the oral cavity were also registered.

- Sialometries As secondary measurements, both unstimulated and stimulated salivary flow rates were assessed in all patients. The unstimulated salivary flow rate was obtained by the spit method every 30 seconds for 15 minutes. Saliva was collected in 20 mL plastic containers, which were pre-weighted (in 0.001 g) using a precision scale. Measurements were expressed as mL/min. Stimulated whole saliva was obtained by chewing a 1 g piece of paraffin wax for six minutes. Saliva collected during the first minute was discarded, and then collected into the container every 30 seconds. Both DMQ and sialometries were always assessed at the same time of day (from 09:00 to 11:00 a.m.) to avoid any circadian variation. Before the evaluation, participants were asked not to eat, drink, smoke or brush their teeth for one hour prior to their appointment at the clinic.Time passed between the last use of the sialogogue and the salivary flow measurements was 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Xerostomia
* Drug consumption
* Antidepressant and antihypertensive agents

Exclusion Criteria:

* Systemic diseases
* Head and neck radiotherapy
* Intake of drugs with high xerostomizing capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gómez-Moreno, Professor, Principal Investigator — Universidad de Granada
Locations (1):
- Dental School, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Malic Acid 1%: Intervention group subjects was the delivery to the patients of a topical sialogogue, containing 1% malic acid, xylitol 10% and fluoride 0.05%(Xeros Dentaid Spray©, Dentaid, Barcelona, Spain).
  Spray was transferred by foreign personnel into identical opaque flasks(without any brand name)labeled A.
  Malic Acid: Oral spray for application into the oral cavity
Period: Overall Study
Arm/Group | Malic Acid 1% | Control
Started | 100 | 85
Completed | 91 | 79
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Malic Acid 1% | Control | Total
Number analyzed (Participants) | 100 | 85 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 85 | 185
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 55 | 123
  Male | 32 | 30 | 62
Region of Enrollment [Number; unit: participants] — Participants were reruited from University of Granada who were attended at dental school
  participants
    Spain | 100 | 85 | 185

OUTCOME MEASURES:

1. Primary Outcome: Dry Mouth Questionnaire (DMQ)
Description: Dry Mouth Questionnaire (DMQ) was used in order to obtain subjective information about the severity of xerostomia before and after treatment with malic acid/placebo.
  Every participant answered an initial questionnaire (DMQ 1) about the symptoms related to oral dryness, before receiving a spray (1% malic acid or placebo). After two weeks of applications, patients had to answer DMQ 1 again as well as an additional questionnaire (DMQ 2) about the efficacy of the sprays. Increased DMQ scores indicate improvement of xerostomia. DMQ 1 was used to assess the initial severity of oral dryness and in particular its impact on oral function: problems when chewing, swallowing, speaking and general impact on daily life.
  DMQ 1 used a 0-to-4 rating scale where 0 = "very dry" and 4 = "not dry at all." After two weeks of treatment, DMQ 1 was repeated and it was included DMQ 2.
  At the end values of DMQ 1 and DMQ 2 were summed
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Malic Acid 1% | Control
Number analyzed (Participants) | 91 | 79
units on a scale | 3.4 (0.6) | 1.4 (0.5)

2. Secondary Outcome: Sialometries
Description: Unstimulated and stimulated salivary flow rates were assessed in all patients. The unstimulated salivary flow rate was obtained by the spit method every 30 seconds for 15 minutes. Saliva was collected in 20 mL plastic containers, which were pre-weighted.
  Stimulated whole saliva was obtained by chewing a 1 g piece of paraffin wax for six minutes. Saliva collected during the first minute was discarded, and then collected into the container every 30 seconds.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Malic Acid 1% | Control
Number analyzed (Participants) | 91 | 79
mL/min
  Unstimulated Salivary Flow rate | 0.17 (0.07) | 0.16 (0.09)
  Stimulated Salivary Flow Rate | 0.93 (0.27) | 0.75 (0.35)

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Malic Acid 1%: Patients treated with Malic Acid 1%
- Control: Patients treated with a placebo
Arm/Group | Malic Acid 1% | Control
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/85
Other Adverse Events (participants affected / at risk) | 0/100 | 0/85

LIMITATIONS AND CAVEATS:
Some of the participants forgot the appointment because the time between phases were of two weeks

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No